CLINICAL TRIAL: NCT01285700
Title: A Single Center, Randomized, Open-label, Multiple-dose Study of the Efficacy and Long-term Safety of rhLAMAN (Recombinant Human Alpha-mannosidase or Lamazym) for the Treatment of Patients With Alpha-mannosidosis.
Brief Title: Dose Finding Study of Recombinant Human Alpha-mannosidase for the Treatment of Patients With Alpha-mannosidosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zymenex A/S (Industry)
Collaborators: European Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rhLAMAN-03; 2010-022085-26 (EudraCT Number)
Record Dates: First submitted 2011-01-25; First posted 2011-01-28 (Estimated); Last update posted 2012-09-26 (Estimated); Status verified 2012-09

CONDITIONS: Alpha Mannosidosis
MeSH Terms: conditions — alpha-Mannosidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lamazym 25 (Active Comparator): 25 U/kg
  Interventions: Drug: Lamazym
- Lamazym 50 (Active Comparator): 50 U/kg
  Interventions: Drug: Lamazym

INTERVENTIONS:
Drug: Lamazym — ERT, infusion weekly
  Other Names: rhLAMAN

SUMMARY:
This is a single-center, open-label, multiple-dose study of the efficacy and long-term safety of Lamazym for the treatment of patients with alpha-mannosidosis.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have a confirmed diagnosis of alpha-Mannosidosis as defined by alpha-mannosidase activity < 10% of normal activity in blood leukocytes
2. The patient must have an age at the time of screening ≥ 5 year and ≤ 21 years
3. The patient must have physical ability to perform 6-minutes walk test (6MWT), 3 minute-stair climb test (3MSCT) and pulmonary lung function test (spirometry, body plethysmography).
4. The patient must have the ability to mentally cooperate in the cognitive and motor function tests
5. The patient must have the ability to hear and follow a request. Hearing aids can be worn.
6. Patient or patient's legally authorized guardian(s) must provide signed, informed consent prior to performing any study-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject)
7. The patient and his/her guardian(s) must have the ability to comply with the protocol

Exclusion Criteria:

1. The patient cannot walk without support.
2. Presence of known chromosomal abnormality and syndromes affecting psychomotor development, other than alpha-Mannosidosis
3. History of bone marrow transplantation
4. Presence of known clinically significant cardiovascular, hepatic, pulmonary or renal disease or other medical conditions that, in the opinion of the Investigator, would preclude participation in the trial
5. Presence of an ECHO with abnormalities within half a year that, in the opinion of the Investigator, would preclude participation in the trial
6. Any other medical condition or serious intercurrent illness, or extenuating circumstance that, in the opinion of the investigator, would preclude participation in the trial
7. Pregnancy
8. Psychosis within the last 3 months

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Reduction of Oligosaccharides in urine | 3 months (interim evaluation) + 6 months
  Efficacy endpoint evaluation as change from baseline

SECONDARY OUTCOMES:
Reduction of Oligosaccharides in serum | 3 months (interim evaluation) + 6 months
  Efficacy endpoint evaluation as change from baseline
Reduction of Oligosaccharides in CSF | 3 months (interim evaluation) + 6 months
  Efficacy endpoint evaluation as change from baseline
The distance walked in 6 minutes | 3 months (interim evaluation) + 6 months
  Efficacy endpoint evaluation as change from baseline
The number of steps climbed in 3 minutes | 3 months (interim evaluation) + 6 months
  Efficacy endpoint evaluation as change from baseline
Pulmonary Function | 3 months (interim evaluation) + 6 months
  Efficacy endpoint evaluation as change from baseline
Adverse events | 1 week
  Safety endpoint assessed weekly throughout the trial
Development of clinically significant changes in vital signs and change in physical examination | 1 week
  Safety endpoint assessed weekly throughout the trial
Development of clinically significant changes in the clinical laboratory parameters (hematology, biochemistry and urinalysis) | 4 weeks
  Safety endpoint assessed every 4th week throughout the trial
Development of rhLAMAN antibodies and neutralizing/inhibitory antibodies | 2 weeks
  Safety endpoint assessed every other week throughout the trial

CONTACTS AND LOCATIONS:
Overall Officials: Allan M. Lund, MD, Principal Investigator — Department of Clinical Genetics, Juliane Marie Centre, Region Hovedstaden, Copenhagen University hospital, Denmark; Jens Fogh, Study Chair — Zymenex A/S
Locations (1):
- Department of Clinical Genetics, Juliane Marie Centre, Copenhagen University Hospital, Blegdamsvej 9, Copenhagen, Denmark